CLINICAL TRIAL: NCT03507179
Title: Retention of Complete Denture Using Rapid Prototyping Versus a Conventional Complete Denture: Cross Over Randomized Control Trial
Brief Title: Retention of Complete Denture Using Rapid Prototyping
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, lina khalaf, teaching assistant, Cairo University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: lina''s protocol
Record Dates: First submitted 2018-04-02; First posted 2018-04-24 (Actual); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Retention of 3D Printed Dentures

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional dentures (Placebo Comparator): a complete denture made through conventional processing technique
  Interventions: Other: conventional dentures
- 3d printed dentures (Active Comparator): a complete denture made through 3D printing
  Interventions: Other: 3d printed denture

INTERVENTIONS:
Other: 3d printed denture — construction of a 3d printed denture through a recent method instead of conventional processing
  Arms: 3d printed dentures
Other: conventional dentures — conventional dentures
  Arms: conventional dentures

SUMMARY:
Nineteen patients will be selected from the clinic following the inclusion and exclusion criteria. Each one of them will receive two dentures. The first denture will be a conventional complete denture while the second denture will be a complete denture made by Rapid prototyping method.

For both groups, a preliminary impression will be made & after pouring the primary impression, self-cured acrylic resin trial denture bases with a wax rim will be constructed on the primary casts for the upper & lower arches for a jaw relation record. A facebow record will be used to mount the upper cast, while the lower cast will be mounted using a centric relation record. Setting of artificial teeth will be performed, then the denture will be tried in patient's mouth. Functional impression will be taken during the try in stage which.

For the first denture, the functional impression will be poured in normal way to obtain the master cast. Then Processing will be done in normal way and the denture will be finished and polished and delivered to the patient.

But for the second denture construction CBCT scanning of the try in with the functional impression will be done to obtain STL file then denture base manufacturing will be done by 3D printing.

For group A and group B Retention will be measured for the upper denture immediately, with a wash out period one month between the two dentures.

DETAILED DESCRIPTION:
Heat processed denture base is the treatment of choice for most of edentulous patients and it is considered as the golden standard and the main comparator for the new techniques. But using Heat Cured Acrylic resin would require many laboratory steps which introduce several errors . Meanwhile, the introduction of rapid prototyping method with high accuracy which eliminates some of the laboratory steps was the reason for choosing it to compare it with the conventional method.

ELIGIBILITY:
Inclusion Criteria:

1. Age ranging from 40-70 years.
2. Cooperative patients.
3. male or female patients

Exclusion Criteria:

1. Pathological changes of residual ridges.
2. Patients with any systemic diseases.
3. Patients with xerostomia.
4. Patients with flabby and flat ridges.
5. Patients with allergy to resins.
6. Patient with sever undercuts, or irregular bony exostosis. -

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2018-05-04 (Estimated); Primary Completion 2018-10-04 (Estimated); Study Completion 2018-11-04 (Estimated)

PRIMARY OUTCOMES:
retention | immediately after denture construction
  We will Determine the geographic center for upper denture base to measure retention then A loop will be attached to each denture base at the position of geographic center using clear self cure acrylic resin and the retention will be measured by applying the forces perpendicular to the denture using Digital Force Meter Each base will be tested 3 times and the average will be calculated. Then the loop will be removed and the denture will finished and polish. Retention will be measured immediately after denture insertion.

IPD SHARING:
Plan to Share IPD: Undecided